CLINICAL TRIAL: NCT06948331
Title: A Pilot Proof of Concept Single-arm Study Using PuraStat Following the Aquablation Procedure to Assess Reduction of Hematuria to Allow for Same Day Discharge
Brief Title: RADA16 for Aquablation Day Case
Acronym: RAD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-00109
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hematuria; Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Hematuria; Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Men Undergoing Aquablation (Experimental): Following the Aquablation procedure for lower urinary tract symptoms (LUTS) due to benign prostatic hyperplasia (BPH), the surgeon will deliver the PuraStat to the prostatic fossa through the cystoscope sheath into the prostate urethra resection bed.
  Interventions: Device: PuraStat

INTERVENTIONS:
Device: PuraStat — Sterile gel composed of synthetic peptide and sterile water; provided as a prefilled syringe. The will be applied to the inside of the prostate to help stop bleeding following Aquablation.

SUMMARY:
This is a pilot proof of concept single-arm study using PuraStat following Aquablation procedure to assess reduction of hematuria to allow for same day discharge.

The primary objective is to assess how PuraStat affects post-operative hematuria following Aquablation.

The secondary objective is to assess the number of patients discharged on the same day based on the hematuria criteria (Grade 0 and Grade I).

ELIGIBILITY:
Inclusion Criteria:

• Any man undergoing Aquablation for LUTS due to BPH

Exclusion Criteria:

• Unwilling to sign consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patients Discharged the Same Day as Aquablation | Day 1 (Operative Visit)

SECONDARY OUTCOMES:
Mean Post-Operation Hematuria Grade | Day 1 (Up to Hour 3 Post-Op)
  The mean hematuria grade noticed 1-3 hours post procedure.
Percentage of Patients who Experience Dysuria during Follow-Up | Up to Week 4 Post-Operation

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kelly, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: chris.kelly@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to chris.kelly@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.